CLINICAL TRIAL: NCT06534190
Title: A Phase II, Open Label, Multi-center Study of 89Zr-DF-Crefmirlimab for CD8 Positron Emission Tomography in Patients With Locally Advanced or Metastatic Solid Tumours
Brief Title: CD8 PET Imaging in Metastatic Solid Tumours
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10353
Record Dates: First submitted 2023-07-13; First posted 2024-08-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Solid Tumor
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD8 PET imaging (Experimental): 89Zr-Df-crefmirlimab will be administered followed by a PET scan 24 hours later. All patients will undergo a 89Zr-Df-crefmirlimab PET scan at baseline and after treatment with the PD-1 antibody. All patients participating in this imaging trial will undergo preferably 2 but at least one tumour biopsy. The biopsy procedure(s) will be performed after the 89Zr-Df-crefmirlimab PET scan at baseline and/or after the 89Zr-Df-crefmirlimab PET on-treatment.
  After the first PET scan and tumour biopsy the patients will start treatment with PD-1 antibody nivolumab or cetrelimab.
  Interventions: Radiation: 89Zr-Df-crefmirlimab PET scan; Drug: Nivolumab; Drug: Cetrelimab; Other: zirconium Zr 89 crefmirlimab berdoxam

INTERVENTIONS:
Radiation: 89Zr-Df-crefmirlimab PET scan — 89Zr-Df-crefmirlimab will be administered followed by a PET scan 24 hours later. All patients will undergo a 89Zr-Df-crefmirlimab PET scan at baseline and after treatment with the PD-1 antibody. All patients participating in this imaging trial will undergo preferably 2 but at least one tumour biopsy. The biopsy procedure(s) will be performed after the 89Zr-Df-crefmirlimab PET scan at baseline and/or after the 89Zr-Df-crefmirlimab PET on-treatment.
  After the first PET scan and tumour biopsy the patients will start treatment with PD-1 antibody nivolumab or cetrelimab.
Drug: Nivolumab — Immunotherapy treatment with Nivolumab
Drug: Cetrelimab — Immunotherapy treatment with cetrelimab
Other: zirconium Zr 89 crefmirlimab berdoxam — 89Zr-Df-crefmirlimab will be administered followed by a PET scan 24 hours later
  Other Names: Zr-89 crefmirlimab berdoxam; 89Zr-Df-crefmirlimab; 89Zr-Df-IAB22M2C

SUMMARY:
This is a multi-center, single-arm trial designed to evaluate the safety and imaging characteristics of 89Zr-Df-crefmirlimab in patients with locally advanced or metastatic solid tumours prior to and during PD-1 antibody therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing informed consent.
2. Patients with histologically confirmed diagnosis of locally advanced or metastatic solid cancer types who, according to the opinion of the principal investigator, based on available clinical data, may benefit from anti-PD1 antibody therapy.
3. Disease progression following first-line therapy or any subsequent treatment line or no superior standard line of therapy available.
4. At least 1 lesion that is accessible per investigator's assessment and eligible for biopsy according to standard clinical care procedures.
5. Measurable disease, as defined by standard RECIST v1.1. Previously irradiated lesions should not be counted as target lesions except for lesions that have progressed after radiotherapy administered at least 3 months earlier.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Life expectancy ≥ 12 weeks.
8. Adequate organ and bone marrow function as defined below:

   1. Hemoglobin ≥9.0 g/dL
   2. Absolute neutrophil count ≥1.0 x 109/L
   3. Absolute lymphocyte count ≥0.75 x 109/L
   4. Platelet count ≥75 x 109/L
   5. Serum creatinine ≤1.5 x upper limit of normal (ULN) or estimated glomerular filtration rate > 30 mL/min/1.73 m2. A 24-hour urine creatinine collection may substitute for the calculated creatinine clearance to meet eligibility criteria.
   6. Adequate hepatic function:

   i. Total bilirubin ≤1.5 x ULN (≤3 x ULN if liver tumour involvement); Patients with Gilbert's syndrome do not need to meet total bilirubin requirements, provided their total bilirubin is unchanged from their baseline. Gilbert's syndrome must be documented appropriately as past medical history.

   ii. Aspartate aminotransferase (AST) ≤2.5 x ULN (≤5 x ULN if liver tumour involvement) iii. Alanine aminotransferase (ALT) ≤2.5 x ULN (≤5 x ULN if liver tumour involvement) iv. Alkaline phosphatase (ALP) ≤2.5 x ULN (≤5 x ULN if liver or bone tumour involvement)
9. Signed informed consent.
10. Willingness and ability to comply with all protocol required procedures.
11. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception (i.e., one that results in a low failure rate (< 1% per year) when used consistently and correctly)).

Exclusion Criteria:

1. Treatment with any approved anti-cancer therapy, investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to 89Zr-Df-crefmirlimab infusion and nivolumab or cetrelimab treatment.
2. Symptomatic, untreated brain metastasis, leptomeningeal disease, or spinal cord compression. Patients are eligible if central nervous system (CNS) metastases are adequately treated and neurologically stable for at least 2 weeks prior to enrollment.
3. Prior ICI treatment, including but not limited to anti-PD1, anti-PD-L1 and anti-CTLA4 therapeutic antibodies.
4. Major surgical procedure other than for diagnosis within 28 days prior to 89Zr-Df-crefmirlimab infusion or anticipation of need for a major surgical procedure during the course of the study.
5. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematous, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis or glomerulonephritis.

   * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for his study.
   * Patients with controlled type I diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
6. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumour necrosis factor agents) within 4 weeks prior to 89Zr-Df-crefmirlimab infusion.

   * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g. a one-time of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the sponsor.
   * The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g. fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
7. Prior allogeneic bone marrow transplantation or solid organ transplant.
8. Active infection with human immunodeficiency virus (HIV), hepatitis B, hepatitis C or tuberculosis infection; or diagnosis of immunodeficiency.

   * Patients will be tested for hepatitis C virus (HCV) and hepatitis B virus (HBV) at screening.
   * Patients with known HIV infection who have controlled infection (undetectable viral load (HIV ribonucleic acid (RNA) polymerase chain reaction (PCR)) and CD4 count above 350 either spontaneously or on a stable antiviral regimen are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
   * Patients with hepatitis B who have a controlled infection (serum HBV deoxyribonucleic acid (DNA) PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA. Patients must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
   * Patients who are HCV antibody positive who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
   * Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
9. Receipt of a live vaccine (including attenuated) within 30 days of planned start of study medication.
10. Evidence of an active infection that requires systemic antibiotics within 2 weeks prior to 89Zr-Df-crefmirlimab infusion.
11. At least 2 weeks recovered from COVID 19 infection, where this infection has to be documented in the case record form.
12. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of 89Zr-Df-crefmirlimab, or that may affect the interpretation of the results or render the patient at high risk from complications.
13. Altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
14. Sponsor employee/member of the clinical site study team and/or his or her immediate family
15. Women with a positive serum chorionic gonadotropin HCG pregnancy test at the screening/baseline visit. Breastfeeding women are also excluded.
16. Women of childbearing potential* and sexually active men who are unwilling to practice highly effective contraception prior to the first dose of study therapy, during the study, and for at least 6 months after the last dose. Highly effective contraceptive measures include:

    * stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening
    * intrauterine device (IUD); intrauterine hormone-releasing system (IUS)
    * bilateral tubal ligation
    * vasectomized partner (provided that the male vasectomized partner is the sole sexual partner of the women of childbearing potential (WOCBP) study participant and that the vasectomized partner has obtained medical assessment of surgical success for the procedure)
    * and/or sexual abstinence.
17. Contraindications for MRI scan
18. Patients who have any splenic disorders, or had splenectomy, that could compromise protocol objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Whole body distribution of 89Zr-Df-crefmirlimab | 2 years
  Evaluate whole body distribution of 89Zr-Df-crefmirlimab in cancer patients prior to and during treatment with an anti-PD-1 antibody by measuring standardized uptake values (SUV) in tumours, healthy tissues and organs.
Pharmacokinetics (PK) of 89Zr-Df-crefmirlimab | 2 years
  Description of pharmacokinetics (PK) of 89Zr-Df-crefmirlimab by measuring standardized uptake value (SUV) on PET scans performed in patients prior to and during treatment with an anti-PD-1 antibody.
Tumour tracer uptake with immune cell CD8 expression | 2 years
  Results of immunohistochemical (IHC) scoring of CD8 expression will be described. These IHC results will be compared with imaging tracer standardized uptake value (SUV) in defined volumes of interest (VOIs) of tumor lesions on the PET scan images.
Changes in tumour volumetry, mpMRI parameters and MRI based texture metrics | 2 years
  DCE-MRI sequences will be evaluated and both semi-quantitative and pharmacokinetic quantitative parameters will be derived using a two-compartmental model.

SECONDARY OUTCOMES:
Incidence, nature, and severity of adverse events (AE) according to NCI-CTCAE v5.0 | Up to 100 days after the last study procedure (treatment discontinuation visit)
  Adverse events will be assessed using the NCI-CTCAE v5.0 criteria, categorizing the severity from Grade 1 (mild) to Grade 5 (death).
correlate mpMRI parameters | 2 years
  correlate mpMRI parameters such as Ktrans derived from DCE-MRI; f, D derived from IVIM-DWI and DDKI and K derived from DK-MRI with tumour and immune cell CD8 expression as well as T cell infiltration
Treatment response with nivolumab or cetrelimab | 2 years
  correlate response to treatment with nivolumab or cetrelimab, according to the RECIST v1.1 and iRECIST criteria with 89Zr-Df-crefmirlimab uptake in tumour lesions.

OTHER OUTCOMES:
89Zr-Df-crefmirlimab uptake with markers of immune infiltrates and other biomarkers for response to ICI therapy | 2 years
  Results of immunohistochemical (IHC) scoring of markers of immune infiltrate other then CD8 expression, such as PDL1, will be described as a semi-quantative score. These IHC results will be compared with imaging tracer standardized uptake value (SUV) in defined volumes of interest (VOIs) of tumor lesions on the PET scan images.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth G.E. de Vries, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (4):
- Netherlands (2):
  - VUMC, Amsterdam
  - University Medical Center Groningen, Groningen
- Vall d'Hebron Institute of Oncology (VHIO) / Vall d'Hebron Institute Research (VHIR), Barcelona, Spain
- University of Cambridge, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided